CLINICAL TRIAL: NCT03764683
Title: A Double-Blind Sequential Parallel Study of Suvorexant (Belsomra) for the Treatment of Bipolar Depression With Insomnia
Brief Title: Suvorexant (Belsomra) for the Treatment of Bipolar Depression With Insomnia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to COVID-19.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P002157
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder; Insomnia
MeSH Terms: conditions — Bipolar Disorder; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: The investigators are proposing the use of SPCD for this study. The Sequential Parallel Comparison Design aims to reduce the impact of high placebo response and decrease sample size. The design has been accepted by and published on by FDA. The SPCD model has two relatively short phases of treatment of equal duration. Only non-responders to placebo (P) during the first phase are included in the analyses of the second phase. Randomization is unbalanced (for example, a 2:3:3 assignment of DD, PP, and PD).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Drug-Drug (Experimental): This arm will receive the active drug in the first and second phase of the study.
  Interventions: Drug: Suvorexant (Belsomra)
- Placebo-Drug (Other): This arm will receive placebo in the first phase of the study and the active drug in the second phase.
  Interventions: Drug: Suvorexant (Belsomra); Drug: Placebo
- Placebo-Placebo (Placebo Comparator): This arm will receive placebo in the first phase and second phase of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant (Belsomra) — Suvorexant (Belsomra) is approved by the U.S. Food and Drug Administration (FDA) to treat insomnia. It has not yet been studied in people with bipolar disorder who have problems sleeping.
  Arms: Drug-Drug; Placebo-Drug
Drug: Placebo — Subjects will take placebo capsules (containing no active substance) identical in appearance to those containing Suvorexant
  Arms: Placebo-Drug; Placebo-Placebo

SUMMARY:
The investigators are doing this research study to find out if suvorexant (Belsomra) can help people with bipolar depression when added to their usual treatment. The investigators also want to find out if suvorexant (Belsomra) is safe to take without causing too many side effects in people with bipolar disorder.

Suvorexant (Belsomra) is approved by the U.S. Food and Drug Administration (FDA) to treat insomnia. It has not yet been studied in people with bipolar disorder who have problems sleeping.

This research study will compare suvorexant (Belsomra) to placebo. The placebo looks exactly like suvorexant (Belsomra), but contains no suvorexant (Belsomra). During this study participants may get a placebo instead of suvorexant (Belsomra). Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

This study has two parts, each lasting 6 weeks. During each part, participants may receive either Belsomra or placebo. Some participants will receive suvorexant for both parts, some will receive placebo for both parts, and others will receive suvorexant during one part and placebo during the other part. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

This study is open to people with bipolar disorder who have trouble sleeping. Bipolar disorder is a brain disorder associated with episodes of mood swings ranging from depressive lows to manic highs.

About 80 subjects will take part in this research study. All subjects will be enrolled at Massachusetts General Hospital (MGH).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 and 75.
2. DSM V diagnosis of Bipolar Disorder Type I and II.
3. Ability to sign the Informed Consent Form.
4. Not taking an antidepressant medication within the past 14 days.
5. Meets criteria for a current major depressive episode as defined and operationalized by the MINI.
6. Patients must have a 10-item MADRS Rating Scale for Depression score ≥ 16 and item 4 (Reduced sleep) score ≥ 4 during the screening phase and at baseline to qualify for inclusion.
7. Scores >15 on the QIDS-SR.
8. Does not meet criteria for current hypomanic or manic episode as defined and operationalized by the MINI 7.0.2.
9. Patients must be stable on their bipolar medications for at least 1 month (4 weeks) prior to screening.

Exclusion Criteria:

1. Unable to sign the Informed Consent Form.
2. Declines to participate.
3. DSM-V diagnosis of Psychosis, Schizophrenia, Schizoaffective Bipolar type.
4. Meets criteria for current hypomanic or manic episode as defined and operationalized by the MINI.
5. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (e.g. oral contraceptives, intrauterine device, barrier methods, or total abstinence from intercourse; Depo Provera is acceptable if it is started 3 months prior to enrollment).
6. Patients who are a serious suicide or homicide risk, suicidal exclusion criteria as follows:

   1. Suicidal ideation associated with actual intent and a method or plan in the past year: "Yes" answers on items 4 or 5 of the C-SSRS
   2. Previous history of suicidal behaviors in the past one year: "Yes" answer (for events that occurred in the past year) to any of the suicidal behavior items of the C-SSRS. (Non-suicidal self-injurious behavior is not included unless in the investigator's judgment it is indicated).
   3. Any lifetime history of serious or recurrent suicidal behavior.
   4. In the investigator's judgment further risk assessment or exclusion due to suicidality is required.
7. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
8. The following DSM-V diagnoses: 1) organic mental disorders; 2) substance use disorders, including alcohol but excluding tobacco, active within the 3 months; 3) schizophrenia; 4) delusional disorder; 5) psychotic disorders not elsewhere classified; 6) schizoaffective disorder; 7) acute bereavement; 9) severe borderline or antisocial personality disorder.

   a. Subjects who have a positive urine drug screen which cannot be explained by prescribed medications, or for which patients do not have a valid prescription for a valid medical reason.
9. Patients meeting criteria for current bipolar mixed episode as defined and operationalized by the MINI.
10. Patients with mood congruent or mood incongruent psychotic features.
11. Clinical or laboratory evidence of hypothyroidism.
12. Patients previously treated with Suvorexant (Belsomra)
13. Patients who have taken an investigational psychotropic drug within the last 60 days.
14. Standard multivitamins with or without minerals will be allowed (with no more than 400 mcg folate) if initiated at least 12 weeks prior to Baseline. Dietary supplements with putative CNS activity will be excluded including SAMe, St. John's Wort, DHEA, Inositol, and Ginko biloba.
15. Previous treatment with the following procedures: ECT, vagus nerve stimulation, or deep brain stimulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality via Pittsburgh Sleep Quality Index (PSQI) | The PSQI will assess change in perceived sleep quality from Week 1 to Week 8 to Week 10 to Week 12 to Week 14.
  The PSQI assesses perceived sleep quality more generally and consists of 7 components: [1] subjective sleep quality (1 item) [2] sleep latency (2 items) [3] sleep duration (1 item) [4] habitual sleep efficiency (3 items) [5] sleep disturbances (9 items) [6] use of sleeping medications (1 item), and [7] daytime dysfunction (2 items).19 items are included in scoring. Five additional items, to be completed by a bed partner, are included in the questionnaire and may be useful for clinical purposes but are not used for scoring.
  The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5"or greater indicates a "poor" sleeper. Lower scores indicate better sleep quality and better outcome. Minimum score is 0, maximum score is 21.
Change in depressive symptoms via the Bipolar Inventory of Symptoms Scale (BISS) | The BISS will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The BISS is a 45-item scale completed by the physician or trained rater, using a structured interview to assess for symptoms of mania and depression (Bowden et al., 2007; Gonzalez et al., 2008). The BISS includes all items from the Montgomery Asberg Depression Rating Scale (MADRS) and the Young Mania Rating Scale (YMRS), plus additional items that are either absent or indirectly addressed in the MADRS and YMRS scales.
  Items are scored from 0 to 4, based on the most recent 7 day period, utilizing information from self report, and family and clinician observation both outside and during the interview. Items are scored both on the basis of frequency and severity. A score of 3, in most cases, also entails behavior that is observable to others. A score of 0 means the symptom is completely absent.
  The Depression subscale of the BISS includes 21 items. Minimum score is 0 and maximum score is 84. Lower scores indicate less severe depressive symptoms and better outcome.
Change in manic symptoms via the Bipolar Inventory of Symptoms Scale (BISS) | The BISS will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The BISS is a 45-item scale completed by the physician or trained rater, using a structured interview to assess for symptoms of mania and depression (Bowden et al., 2007; Gonzalez et al., 2008). The BISS includes all items from the Montgomery Asberg Depression Rating Scale (MADRS) and the Young Mania Rating Scale (YMRS), plus additional items that are either absent or indirectly addressed in the MADRS and YMRS scales.
  Items are scored from 0 to 4, based on the most recent 7 day period, utilizing information from self report, and family and clinician observation both outside and during the interview. Items are scored both on the basis of frequency and severity. A score of 3, in most cases, also entails behavior that is observable to others. A score of 0 means the symptom is completely absent.
  The Mania subscale of the BISS includes 21 items. Minimum score is 0 and maximum score is 84. Lower scores indicate less severe manic symptoms and better outcome.
Change in psychosocial functioning via Quality of Life Satisfaction Questionnaire (Q-LES-Q) | The Q-LES-Q will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The Q-LES-Q is a patient-administered instrument, which has a "long" and "short" form (Endicott, 1993). The "long" form asks questions in 8 modules of 6-16 questions each, about physical health/activities, general feelings of well-being and relaxation, function at work, household duties, school or course work, leisure activities, social relations, and general activities over the past week. Patients will be administered the "long form" version.

SECONDARY OUTCOMES:
Change in insomnia measured via Insomnia Severity Index (ISI) | This will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The ISI measures the subjective symptoms and consequences of difficulties initiating and maintaining sleep and self-perception of insomnia symptoms as well as the degree of concerns or distress caused by those symptoms. This scale includes 7 items, each scored on a 0-4 scale. Items are summed to produce a total score with a maximum of 28 and minimum of 0. Change in total score (sum of scores from 7 items) is used for study outcome Lower scores indicate less severe insomnia symptoms and better outcome.
Change in bipolar symptom severity via Clinical Global Impressions - Severity (CGI-S) | This will be administered at Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The CGI-S is a rating of severity of the disorder since beginning of the study. This instrument is completed by the clinician based on assessment of the patient's clinical status. Based on history and scores on other instruments, the clinician assesses the current condition of the patient on a scale of 1-7 (1 being normal, and 7 being among the most severely ill patients). A decrease in CGI-S indicates less severe bipolar symptoms and better outcome.
Change in suicidal ideation score on The Columbia Suicide Severity Rating Scale (C-SSRS) | This will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior to assess severity of and to track suicidal events throughout any treatment.
  It includes categories: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide. Suicidal Ideation Score is a numerical score calculated from the above categories, with some categories scored on a 1-5 scale and others on a 0-5 scale. Change in total score (sum of scores from 5 categories; max. score=25, min. score=3) is used for study outcome. Lower Suicidal Ideation Score indicates less severe suicidal ideation and better outcome.
Change in functioning via MGH Cognitive and Physical Functioning Questionnaire (MGH-CPFQ) | This will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The MGH-CPFQ is a brief scale used to measure cognitive and executive dysfunction in mood and anxiety disorders (Fava, Iosifescu, Pedrelli, & Baer, 2009). The MGH-CPFQ will allow for assessment of symptoms such as fatigue, apathy, and neuropsychological functioning.The scale includes 7 items, each scored on a 1-6 scale with a lower score indicating less severe functional impairment. Change in total score (sum of scores from 7 items) is used for study outcome, with a lower score indicating better outcome. Minimum total score is 7 and maximum total score is 42.
Change in depressive symptoms via Quick Inventory of Depression Symptomatology-Self Report (QIDS-SR) | This will be administered at Screen visit, Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 14.
  The QIDS-SR is the self-rated equivalent to the QIDS-CR and has excellent agreement with the clinician rated scale (Rush et al., 2003; 2005). The QIDS-SR will allow assessment of patient perception of illness and improvement. This measure includes 16 items, each scored on a 0-3 scale with 0 indicating less severe depressive symptoms. Change in total score (sum of scores from 16 items) is used for study outcome, with a lower score indicating better outcome. Minimum total score is 0 and maximum total score is 48.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Kinrys, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.